CLINICAL TRIAL: NCT03402425
Title: The Diagnostic Value of 18F-FET PET/MRI for CNS Tumors in Children and Adolescents
Acronym: BUF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Børnecancerfonden (Other)
Responsible Party: Principal Investigator, Lisbeth Marner, MD, PhD, DMSc, Staff Specialist, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 327-15
Record Dates: First submitted 2017-05-01; First posted 2018-01-18 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Positron-Emission Tomography; Brain Neoplasms, Childhood
Keywords: FET; PET/MRI; child
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: We aim to include all patients that fullfil the inclusion criteria.
Masking Description: The result of the PET scan is masked until a treatment plan for the patient has been decided by the treatment responsible clinicians based on the MRI findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All included patients (Experimental): A 18F-FET PET scan is performed
  Interventions: Diagnostic Test: 18F-FET PET

INTERVENTIONS:
Diagnostic Test: 18F-FET PET — Patient are investigated with an 18F-FET PET

SUMMARY:
To investigate the diagnostic value of 18F-FET PET/MRI instead of MRI alone, children and adolescents with tumor in brain or spinal cord are included and scanned primarily at our hybrid PET/MRI using the amino acid analog 18F-FET. The scans are performed at primary diagnosis, before radiation therapy, before and after operation, when relapse is suspected and three or six months after initiation of chemotherapy.

DETAILED DESCRIPTION:
Background. Tumors in the brain and spinal cord are among the most common causes of death and disability by cancer in children and adolescents. MRI is used for primary diagnosis as well as follow-up but is often challenged by tissue changes caused by the treatment. The amino acid analog 18F-FET is used increasingly in adults to delineate tumor and discriminate tumor from treatment effects. A hybrid PET/MRI scanner enables the simultaneous imaging with PET and MRI, which is important in especially the younger children needing anaesthesia to cooperate to the procedure.

Aim The aim of the study is to compare diagnostics using MRI alone with 18F-FET PET/MRI (or sequential MRI and PET) in children and adolescents diagnosed with a central nervous system (CNS) tumor before the age of 18 years. The scans will be performed at primary diagnosis/before operation/biopsy, within 72 hours after operation, planning radiation therapy, evaluation of treatment effect, when relapse is suspected.

Exclusion criteria are MRI contraindications, pregnancy, or a syndrome with increased sensitivity to radiation.

The investigators wish to evaluate which cases and for which tumor types, 18F-FET PET/MRI will increase sensitivity and specificity of diagnosing CNS tumors.

Side effects The side effects are mainly the side effect from the MRI with venous puncture, the MRI contrast leading that can lead to shortlived nausea or headache, fasting for 6 hours and the radioactivity exposure of 4.2 mSv (1,4 times the early background radiation) for each scan procedure. The maximal number of scans in the project is 3, 6 or 10 depending on the diagnosis.

Data Analysis The correlation between 18F-FET uptake in tumor and tumor grading (obtained from operation/biopsy) will be investigated.

When relapse is suspected, sensitivity and specificity for recurrence/progression for MRI alone versus PET/MRI will be compared.

It will be analysed if the addition of PET influences the diagnosis/chosen treatment. A major impact of 6% will be regarded significant.

The prognostic value of 18F-FET uptake after treatment will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of newly diagnosed CNS tumor, recurrence or radiation therapy planning
* age <18 years at first CT/MRI suggesting CNS tumor
* written informed consent from parents (age < 18 years) or the patient (age >18 years)

Exclusion Criteria:

* contraindications for MRI (e.g. metal implants)
* pregnancy
* known syndrome with increased sensitivity to radiation (e.g. Gorlin or Ataxia Telangiectasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-02-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of treatment | up to 3 months
  The treatment plan is changed based on the PET findings

SECONDARY OUTCOMES:
Sensitivity and specificity | up to 3 months
  The sensitivity and specificity of PET/MRI is compared to MRI alone. The gold standard is clinical follow-up.
Recurrence free survival time | at least one year
  Comparison of PET better than MRI can predict the time before progression or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Marner, MD PhD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital Rigshospitalet, Copenhagen, Copenhagen O, Denmark

IPD SHARING:
Plan to Share IPD: No